CLINICAL TRIAL: NCT05638815
Title: An Observational Study to Explore the Role of Alpha-Synuclein-related Biomarkers in the Diagnosis and Disease Evaluation of Parkinson's Disease and Other Synucleinopathies
Brief Title: An Observational Study of Parkinson's Disease and Other Synucleinopathies (EASE-PD)
Acronym: EASE-PD
Status: Completed | Type: Observational
Sponsor: SciNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: SNP704
Record Dates: First submitted 2022-03-22; First posted 2022-12-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Parkinson's Disease; Multiple System Atrophy
Keywords: α-synuclein; synucleinopathies; Parkinson's Disease; Multiple System Atrophy
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Parkinson Disease 4, Autosomal Dominant Lewy Body; Synucleinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's Disease (PD)
- Multiple System Atrophy (MSA)
- Health volunteers

SUMMARY:
The study is a multi-center, observational study to evaluate the feasibility of α-synuclein-related biomarkers and imaging data in the disease diagnosis and prognosis evaluation in Synucleinopathies and healthy subjects.

DETAILED DESCRIPTION:
In the study, a total number of no more than 100 subjects are planned to be enrolled.

Subjects who are eligible for enrollment will be enrolled in the study after signing the informed consent form (ICF) and undergo 3 visits, including the baseline visit (the day of first blood sample collection), visit 1 (day 183 post-enrollment), and visit 2 (day 366 post-enrollment).

ELIGIBILITY:
Inclusion Criteria:

* PD subjects must meet the following criteria to be eligible:

  1. Age ≥ 40 years old, regardless of gender;
  2. Primary PD is diagnosed according to MDS Clinical Diagnostic Criteria for Parkinson's Disease of the International Movement Disorders Association (MDS) in 2015 and the Diagnostic Criteria of Parkinson's Disease in China in 2016;
  3. Hohen & Yahr stage 1-3;
  4. Receive standard treatment for at least 4 weeks before the screening visit (standard treatment is listed in the Chinese Guidelines for the Treatment of Parkinson's Disease (Fourth Edition));
  5. The subject or his/her legal representative is able to understand the content of the informed consent and provide a signed ICF.
* MSA subjects must meet the following criteria to be eligible:

  1. Age ≥ 40 years old, regardless of gender;
  2. Patients with probable and possible MSA are diagnosed according to the Second Consensus Statement on the Diagnosis of Multiple System Atrophy and the Chinese Expert Consensus on the Diagnostic Criteria of Multiple System Atrophy in 2018;
  3. The subject or his/her legal representative is able to understand the content of the informed consent and provide a signed ICF.
* Healthy subjects must meet the following criteria to be eligible:

  1. Age ≥ 40 years old, regardless of gender;
  2. Volunteers who are in good health for their age as determined by clinical examination at the time of screening and who are free from dyskinesia as determined by a complete neurological assessment and from serious systemic disease as determined by a complete history;
  3. Be able to understand the content of informed consent and agree to sign ICF.

Exclusion Criteria:

* Excluded if any of the following criteria is met:

  1. Secondary Parkinsonism due to infection, vascular, drugs, poisons, trauma and other causes;
  2. Malignant neoplasm (except basal or squamous cell skin cancer) diagnosed within the last 5 years;
  3. Those with a known mental illness or substance abuse that will cause them to be unable to cooperate;
  4. Patients with severe depression or suicidal behavior (including active attempt, interrupted attempt or attempted attempt) or suicidal thoughts in the past 6 months according to the clinical judgment of the investigator;
  5. Pregnant or lactating women;
  6. Prior treatment with drugs targeting α-synuclein;
  7. Received an investigational drug or device within the previous 4 weeks;
  8. The results of laboratory examination and serological virological examination are not suitable for enrollment according to the judgment of the investigator;
  9. Other conditions judged by the investigator as not suitable for inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: included in the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the difference of α-synuclein-related biomarkers between patients and healthy subjects | 12 months

SECONDARY OUTCOMES:
Attempt to evaluate the correlation between α-synuclein and disease progression by comparing α-synuclein levels at baseline | 6 months, and 12 months
To evaluate the differences of imaging-related indicators in PD, MSA, and their correlation with the disease by brain positron emission tomography (PET) | 12 months
To evaluate the correlation between α-synuclein levels and imaging data. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shengdi Chen, MD,PHD, Principal Investigator — Neurology Department in Ruijin Hospital Shanghai JiaoTong University School of Medicine
Locations (4):
- China (4):
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SciNeuro official website — https://www.scineuro.com/